CLINICAL TRIAL: NCT07309185
Title: Adebrelimab Combined With Famitinib Malate and Irinotecan Versus Irinotecan in Patients With Advanced Gastric Cancer After Failure of First-Line Therapy: A Randomized, Controlled, Exploratory Clinical Study
Brief Title: Adebrelimab Combined With Famitinib and Irinotecan in Advanced Gastric Cancer After Failure of First-Line Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Tumor Hospital (Other)
Responsible Party: Principal Investigator, Xiuping Ding, Prof., Shandong Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-018
Record Dates: First submitted 2025-12-11; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stomach Neoplasms
Keywords: Immune checkpoint inhibitors; Adebrelimab Injection; Famitinib; Second line treatment for advanced
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Adebrelimab Injection: 1200mg, i.v.gtt, d1, Malic acid Famitinib: 20mg, po, d1-21. Irinotecan: 125mg/m2, i.v.gtt, d1, 8. Once every 3 weeks, continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
  Interventions: Drug: Adebrelimab; Drug: Irinotecan; Drug: Malic acid Famitinib
- Group 2 (Active Comparator): Irinotecan: 125mg/m2, i.v.gtt, d1, 8. Once every 3 weeks, continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab Injection: 1200mg, i.v.gtt, d1,
  Once every 3 weeks, continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
  Arms: Group 1
Drug: Irinotecan — Irinotecan: 125mg/m2, i.v.gtt, d1, 8. Once every 3 weeks, continue medication until disease progression, toxicity intolerance, initiation of new anti-tumor treatment, withdrawal of knowledge, or continuous medication for at least 2 years.
Drug: Malic acid Famitinib — Malic acid Famitinib: 20mg, po, d1-21.
  Arms: Group 1

SUMMARY:
This study employs a randomized, controlled, exploratory clinical trial design, with a planned enrollment of 66 patients who have previously failed systemic chemotherapy for recurrent/metastatic gastric cancer,

DETAILED DESCRIPTION:
Among these, 6 cases were in the safety run-in period, receiving treatment with Adeberlimab combined with Famitinib and Irinotecan. The safety during the first 3 months of medication was observed to determine whether DLT (Dose-Limiting Toxicity) occurred within the treatment cycle. If ≤ 2 subjects experienced DLT, the study would proceed to the extension treatment phase; if > 2 subjects experienced DLT, the study would be terminated.

DLT is defined as the occurrence of any of the following drug-related events during the first treatment cycle: grade 4 hematologic toxicity; grade 3 neutropenia with fever; grade 3 thrombocytopenia with bleeding; or any other grade 3 non-hematologic toxicity (excluding alopecia).

After the safety importation period, patients will enter the extended treatment phase, with an additional 60 cases to be enrolled and randomly assigned in a 1:1 ratio to either the experimental group or the control group.

The experimental group received treatment with Adeberlimab combined with famitinib maleate and irinotecan until disease progression, intolerable adverse reactions, or death.

The control group received irinotecan treatment until disease progression, unacceptable toxicity, or death.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with advanced gastric adenocarcinoma or gastroesophageal junction adenocarcinoma diagnosed by histology or cytology;
* 2. Patients who have previously failed first-line treatment including systemic chemotherapy and immune checkpoint inhibitors, and have maintained first-line use of immune checkpoint inhibitors for at least 3 months;
* 3. According to the evaluation criteria for solid tumor efficacy 1.1 (RECIST v1.1), there should be at least one measurable lesion that has not received local treatment such as radiotherapy (lesions located within the previously irradiated area can also be selected as target lesions if progression is confirmed);
* 4. ECOG score: 0-1 point;
* 5. Expected survival period ≥ 12 weeks;
* 6. The main organ functions well and the laboratory test data meets the following standards: (1) Blood routine: absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal laboratory values in the research center), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90g/L; (2) Liver function: serum total bilirubin ≤ 1.5 times the upper limit of the standard value (ULN), AST and ALT ≤ 2.5 times ULN. If the patient has liver metastasis, this standard is ≤ 5 times ULN; (3) Renal function: CrCl ≥ 60 ml/min/1.73 m2 (calculated according to the Cockcroft Gault formula);
* 7. Female subjects with fertility, as well as male subjects with partners who are fertility women, are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period, at least 6 months after the last use of Adebrelimab, and at least 6 months after the last use of chemotherapy;
* 8. Voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* 1. History of gastrointestinal perforation and/or fistula within 6 months prior to the first use of medication;
* 2. There is uncontrollable pleural effusion, pericardial effusion, or peritoneal effusion that requires repeated drainage;
* 3. History of allergies to any component of Adebrelimab in the past;
* 4. Have received any of the following treatments:

  1. Received any other investigational drug within 4 weeks prior to the first use of the investigational drug or had a half-life of no more than 5 from the last investigational drug;
  2. Simultaneously enrolled in another clinical study, unless it is an observational (non interventional) clinical study or an interventional clinical study follow-up;
  3. Received anti-tumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization) within 2 weeks prior to the first use of the investigational drug;
  4. Subjects who need to receive corticosteroids (equivalent to>10mg prednisone per day) within 2 weeks prior to the first use of the study drug. Allow the use of hormones for routine chemotherapy pretreatment without the need for dose adjustment. Other special circumstances require communication with the researcher. In the absence of active autoimmune diseases, inhalation or local use of steroids and corticosteroids with a dosage greater than 10mg/day of prednisone efficacy dose are allowed as substitutes for adrenal cortex hormones;
  5. Individuals who have received anti-tumor vaccines or have received live vaccines within 4 weeks prior to the first administration of the study drug;
  6. Having undergone major surgery or suffered severe trauma within 4 weeks prior to the first use of the investigational drug;
  7. Patients who have received previous treatment with paclitaxel drugs;
* 5. The toxicity of previous anti-tumor treatments has not recovered to ≤ CTCAE 5.0 Grade 1 (excluding hair loss) or the level specified in the inclusion/exclusion criteria;
* 6. Patients with active central nervous system metastases;
* 7. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to the above diseases or syndromes); Excluding childhood asthma/allergies with vitiligo or those who have already recovered, patients who do not require any intervention in adulthood; Autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin;
* 8. Have a history of immune deficiency, including HIV test positive, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation, or active hepatitis (hepatitis B reference: HBV DNA test value exceeds 500 IU/ml or 2500 copies/mL);
* 9. The subject has uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or above heart failure; (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within one year; (4) Clinically significant supraventricular or ventricular arrhythmias that have not been clinically intervened or are still poorly controlled after clinical intervention;
* 10. Within 4 weeks prior to the first use of the investigational drug, there has been a severe infection (CTCAE 5.0>grade 2), such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc; Baseline chest imaging examination suggests the presence of active pulmonary inflammation, symptoms and signs of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except for prophylactic use of antibiotics;
* 11. History of interstitial lung disease (excluding history of radiation pneumonia and non infectious pneumonia that have not been treated with steroids);
* 12. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within the past year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than one year ago but without formal treatment;
* 13. Diagnosed with any other malignant tumor within 5 years prior to the first use of the investigational drug, except for malignant tumors with low-risk metastasis and mortality risk (5-year survival rate>90%), such as basal cell or squamous cell carcinoma or cervical carcinoma in situ that have been adequately treated;
* 14. Pregnant or lactating women;
* 15. According to the researcher's assessment, there may be other factors that could force the subject to terminate the study midway, such as having other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
PFS | The longest follow-up period from the patient's enrollment to disease progression or death from any cause is 2 years
  Progression free survival

SECONDARY OUTCOMES:
mOS | The longest follow-up period from the patient's enrollment to death from any cause is 2 years
  median survival time
DCR | The longest follow-up period from enrollment to the first efficacy evaluation is 3 months
  Disease Control Rate
safety：Record the incidence rate of all adverse events | From enrollment until 90 days after the last dose of medication
  Record the incidence rate of all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bo Liu, Professor, Principal Investigator — Shandong First Medical University Affiliated Cancer Hospital
Locations (1):
- Shandong First Medical University Affiliated Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No